CLINICAL TRIAL: NCT01272726
Title: Influence of Education on Acceptance of Treatment for Attention Deficit Hyperactivity Disorder (ADHD) Among Women
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Principal Investigator, Tammy Jung, Regulatory Specialist, Avera McKennan Hospital & University Health Center
Other Study IDs: ARI-1260-ADHD
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Educational Status; Mental Health

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ADHD: Women with symptoms of ADHD. Women who either think they may have ADHD or have been previously diagnosed with ADHD but have not been treated for it.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Education on the genetics of ADHD and treatment options for ADHD
  Other Names: Attention Deficit Hyperactivity Disorder; Hyperactivity Disorder; Attention Deficit Disorder; Mental Health

SUMMARY:
The goal of this research study is to measure what percentage of women who suspect they have symptoms of ADHD will go on to be diagnosed with ADHD using accepted practice standards. The study will also evaluate the influence education on the genetics of ADHD has on a woman in her deciding to receive behavioral health treatment for ADHD.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) affects approximately 10-12% of school-aged children in the United States, making it one of the most common psychiatric disorders in children. It is characterized as inattention and hyperactivity-impulsivity, which has persisted for at least 6 months to a degree that is maladaptive and inconsistent with developmental level (DSM-IV-TR). ADHD is a non-fluctuating illness unlike many other psychiatric co-morbid conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be females, 18 through 59 years of age
* Subjects must think they have ADHD or have been previously diagnosed with ADHD but may not have received any treatment for ADHD
* Subjects must be able to participate in the informed consent process and give their written consent to participate in the study

Exclusion Criteria:

* Subjects who have been treated (at any time) for ADHD will be excluded from the study
* Potential subjects consuming greater than 21 units of alcohol (1 unit=12.0 ounces beer, 1.5 ounces hard liquor or 5.0 ounces wine) a week will be excluded from the study
* Potential subjects currently experiencing suicidal ideation or who have been hospitalized within the past six months for suicidal ideation will be excluded from the study

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in and around the Sioux Falls area.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine if offering relative risk genotyping for ADHD, and educating around the genetic and environmental contributions to ADHD, may lead to greater health care acceptance in women who struggle with ADHD. | 24 hours

SECONDARY OUTCOMES:
To determine if women who think they have ADHD actually have ADHD. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Soundy, MD, Principal Investigator — Avera McKennan Hospital & University Health Center; Kent Andre, MD, Principal Investigator — Avera McKennan Hospital & University Health Center; Nicole Christensen, MD, Principal Investigator — Avera McKennan Hospital & University Health Center; Gareth Davies, PhD, Study Chair — Avera Institute of Human Behavioral Genetics
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Murphy KR, Adler LA. Assessing attention-deficit/hyperactivity disorder in adults: focus on rating scales. J Clin Psychiatry. 2004;65 Suppl 3:12-7. PMID 15046530
- [Background] Barr CL, Feng Y, Wigg K, Bloom S, Roberts W, Malone M, Schachar R, Tannock R, Kennedy JL. Identification of DNA variants in the SNAP-25 gene and linkage study of these polymorphisms and attention-deficit hyperactivity disorder. Mol Psychiatry. 2000 Jul;5(4):405-9. doi: 10.1038/sj.mp.4000733. PMID 10889551
- [Background] Biederman J, Faraone SV, Keenan K, Knee D, Tsuang MT. Family-genetic and psychosocial risk factors in DSM-III attention deficit disorder. J Am Acad Child Adolesc Psychiatry. 1990 Jul;29(4):526-33. doi: 10.1097/00004583-199007000-00004. PMID 2387786
- [Background] Biederman J, Milberger S, Faraone SV, Kiely K, Guite J, Mick E, Ablon S, Warburton R, Reed E. Family-environment risk factors for attention-deficit hyperactivity disorder. A test of Rutter's indicators of adversity. Arch Gen Psychiatry. 1995 Jun;52(6):464-70. doi: 10.1001/archpsyc.1995.03950180050007. PMID 7771916
- [Background] Faraone SV, Doyle AE. The nature and heritability of attention-deficit/hyperactivity disorder. Child Adolesc Psychiatr Clin N Am. 2001 Apr;10(2):299-316, viii-ix. PMID 11351800
- [Background] Smalley SL, McGough JJ, Del'Homme M, NewDelman J, Gordon E, Kim T, Liu A, McCracken JT. Familial clustering of symptoms and disruptive behaviors in multiplex families with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2000 Sep;39(9):1135-43. doi: 10.1097/00004583-200009000-00013. PMID 10986810